CLINICAL TRIAL: NCT03204422
Title: The Exploratory and Validation Study of Estimation Method of 24-hour Urinary Sodium Excretion by Using Spot Urine for Chinese Children and Adults
Brief Title: Estimation Method of 24-hour Urinary Sodium Excretion by Using Spot Urine for Chinese Population
Status: Completed | Type: Observational
Sponsor: Beijing Children's Hospital (Other)
Collaborators: Capital Medical University (Other)
Responsible Party: Principal Investigator, Yaguang Peng, research assistant, Beijing Children's Hospital
Other Study IDs: 17JL85
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Urinary Sodium Excretion; Salt Intakes
Keywords: urinary sodium excretion; 24-hout urine; salt intakes; hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — the 24-h urine sample and the spot urine samples will be required collected and be retained.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children's group: no intervention. participants, whose age was 5 to 18 years, were enrolled in Children's group.
  Interventions: Other: No intervention
- Adults group: no intervention. participants, whose age was over 18 years, were enrolled in Adults group.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — no any other intervention

SUMMARY:
The accurate evaluation of daily salt or sodium intake is difficult to implement in clinical practice and large epidemiological studies. 24-h urinary sodium excretion (USE) is considered the gold standard, but is expensive and has a high participant burden. To further explore the association between 24-h USE and spot urines in Chinese population, it was proposed that using collected multiple spot urine samples could be estimated for 24-h USE in Chinese children and adults.

DETAILED DESCRIPTION:
Specific Aims

1. To collect multiple spot urine samples and a 24-h urine sample in a population of Chinese Children and adults. All participants will collect a spot urine in separate jugs during the 24-h period, recording every urination time.
2. Validate previous finding that 24-h USE is estimated inaccurately by using only the second morning void.
3. Explore a statistical formula to estimate 24-h USE by multi-time spot urine. The study plan to enroll 200 children and 100 adults to collect a whole 24-h urine spot by spot continuously. After a laboratory examination of sodium concentration from both spot urine samples and 24-h urine sample, the exploratory estimation using multi-spot urine to assess 24-h urinary sodium excretion will analyzed statistically. The validation for the estimation method will be conducted in Chinese population as well.

Urine sodium and potassium concentration in each urine specimen will be determined by ion selective electrode methods and creatinine using enzymatic methods.The model established by using linear model step by step. And the validation analysis conducted through correlation analysis, bias distribution, residual analysis and Bland-Altman plot to assess accuracy. All statistics analysis will be conducted using Statistical Analysis System software version 9.4.

ELIGIBILITY:
Inclusion Criteria:

* Aged 5-60 years
* Provide written informed consent
* Without any renal diseases or conditions which could affect renal function

Exclusion Criteria:

* Pregnant
* Taking diuretic medicine or pharmaceutical using patients, e.g. some hypertension or heart diseases patients
* Cancer patients or some other severe patient

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The children participants will be childrens from children's health care center and some inhospital patients from ophthalmology and orthopaedics ward in Beijing Children's Hospital.
  The adult participants will be residents from community.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
urinary sodium excretion concentration | day 1
  the concentration measured by laboratory examination for the 24 hour urine sample and spot urine samples

CONTACTS AND LOCATIONS:
Overall Officials: Yaguang Peng, PhD, Principal Investigator — Beijing Children's Hospital
Locations (1):
- Beijing Children's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No